CLINICAL TRIAL: NCT01623609
Title: A Phase I, Randomised, Open-label, 3 Way Cross-over Study in Healthy Volunteers to Demonstrate the Bioequivalence of the Naloxegol 25 mg Commercial and Phase III Formulations and to Assess the Effect of Food Administration on the Pharmacokinetics of the Commercial Formulation.
Brief Title: Open Label, Healthy Volunteers, Bioequivalence Study With Naloxegol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00018
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Opioid Induced Constipation
Keywords: Phase 1; Healthy volunteers; Naloxegol; Bioequivalence
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Naloxol IR tablet 25 mg (naloxegol oxalate) commercial formulation under fasted conditions
  Interventions: Drug: Naloxegol
- B (Experimental): Naloxol IR tablet 25 mg (naloxegol oxalate) commercial formulation under fed conditions
  Interventions: Drug: Naloxegol
- C (Experimental): Naloxegol film-coated IR tablet 25 mg Phase III formulation under fasted conditions
  Interventions: Drug: Naloxegol

INTERVENTIONS:
Drug: Naloxegol — Naloxol IR tablet 25 mg (naloxegol oxalate) commercial formulation
  Arms: A; B
Drug: Naloxegol — Naloxegol film-coated Phase III formulation 25 mg film-coated IR tablet
  Arms: C

SUMMARY:
The purpose of this study is to demonstrate the Bioequivalence, assess food administration on the Pharmacokinetics with naloxegol.

DETAILED DESCRIPTION:
A Phase I, Randomised, Open-label, 3 way Cross-over Study in Healthy Volunteers to Demonstrate the Bioequivalence of the Naloxegol 25 mg Commercial and Phase III Formulations and to Assess the Effect of Food Administration on the Pharmacokinetics of the Commercial Formulation.

ELIGIBILITY:
Inclusion Criteria:

* Female non-pregnant, non-lactating.
* Volunteers with suitable veins for cannulation or repeated venipuncture.
* Male healthy volunteers should be willing to use barrier contraception ie, condoms, from the first day of dosing until 3 months after dosing with the investigational product.
* The female partner should use contraception during this period.

Exclusion Criteria:

* History of any clinically significant disease or disorder.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product.
* Volunteers who have smoked or used nicotine products within the previous 3 months from the date of screening.
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results as judged by the Investigator .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic (PK) profile for naloxegol in terms of maximum observed plasma concentration (Cmax) and area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC) for each treatment period. | Predose,0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, clinical laboratory assessments , vital signs (blood pressure and pulse rate), physical examinations, electrocardiograms, and Columbia-Suicide Severity Rating scale (CSSRS) | From baseline day 1 through to Follow-up (Maximum 40 days)
Description of the pharmacokinetic(PK) profile for naloxegol in terms of time to Cmax (tmax), terminal half-life (t1/2λz), terminal rate constant (λz). For each treatment period | Predose,0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours
Description of the pharmacokinetic (PK) profile for naloxegol in terms of area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-t)].For each treatment period | Predose,0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours
Description of the pharmacokinetic (PK) profile for naloxegol in terms of area under the plasma concentration-time curve from time zero to 24 hours [AUC(0-24)], apparent oral clearance from plasma (CL/F).For each treatment period | Predose,0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours
Description of the pharmacokinetic (PK) profile for naloxegol in terms of apparent volume of distribution during the terminal phase (Vz/F)For each treatment period | Predose,0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — Astrazeneca Wilmington, US; Arpeat Kaviya, MBCHB, MRCP, Principal Investigator — Quintiles London UK; Bo Fransson, MD, Study Chair — Astrazeneca Sodertalje Sweden
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: Clinical_Study_Report_Synopsis_D3820C00018 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1397&filename=Clinical_Study_Report_Synopsis_D3820C00018.pdf